CLINICAL TRIAL: NCT05214859
Title: Enhancing Mother-Child Ties and Psychosocial Wellness Through Arts: A Mixed Methods Study on Dyadic Expressive Arts-based Intervention for Children With Intellectual Disability and Their Mothers
Brief Title: Enhancing Mother-Child Ties and Psychosocial Wellness Through Arts Among Children With Intellectual Disability and Their Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Chi Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA200329
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intellectual Disability; Mother-Child Relations
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Due to the nature of this trial, neither the staff, participants, nor care provider can be masked to allocation. The data analyst will be blinded during the data analysis process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive Dyadic Expressive Arts Group Therapy as an intervention.
  Interventions: Behavioral: The Dyadic Expressive Arts Group Therapy
- The Treatment-as-usual Waitlist Control Group (No Intervention): Participants in the control group will continue their routine healthcare and social services. Upon completion of the 8-month study period, participants will be invited to a similar intervention group program.

INTERVENTIONS:
Behavioral: The Dyadic Expressive Arts Group Therapy — This therapy utilizes different art modalities, such as visual art, music, movement, dance, drama, and writing, as therapeutic means. With multiple sensory stimulations from different art forms, the therapy facilitates communication, expression, perception, and interactions. The therapy consists of 8 weekly 90 minutes sessions, with 3-4 mother-child dyads in each therapy group. Each session will follow the basic structure of Expressive Arts Therapy, including check-in, warm-up, core art-making, sharing, and closure. The following themes related to the mother-child relationship will be included, such as communication, relationship, expression, empathy, interaction, love, gratitude, and connection.
  Arms: Intervention

SUMMARY:
The caregiving of children with intellectual disability (ID) is intensive and challenging. Caregivers, particularly mothers, are left in a vulnerable and stressful condition. Children with ID may experience difficulties in expressing emotions and may have behavioral or emotional problems. These difficulties impose extra challenges for the parents to understand and interact with their children with ID. Existing intervention programs for families having children with ID primarily focus on problem-and-emotion-focused measures. While strategies focusing on improving parent-child relationships, mother-child communication, and wellness of the dyads are limited.

Expressive arts-based intervention (EXAT) adopts multiple art modalities for achieving therapeutic goals. It can bypass verbal expression and complicated cognitive processing during interactions, and it is also safe, engaging, enjoyable, and empowering. While existing evidence supports the use of arts-based intervention on children and their parents, there is a limited understanding of the application of dyadic EXAT on the mother-child relationship and their wellness.

The main objective of this study is to evaluate the effectiveness of the dyadic Expressive Arts-based Intervention (EXAT) on the psychosocial well-being of mother-child dyads. Primary outcomes include parent-child relationship, parenting stress, and caregiver burnout; secondary outcomes include mother's affect and quality of life; child's mood, emotional expression, behavioral and emotional problems.

This study adopts a mixed-methods design with quantitative, qualitative, and art-based assessment methods. This study is a randomized controlled trial, running for 3 years for evaluating the effectiveness of the dyadic Expressive Arts-based Intervention (EXAT). 154 Chinese mother-child dyads will be randomized into (i) a dyadic EXAT group or (ii) a treatment-as-usual waitlist control group.

Quantitative analysis will be adopted to investigate the effectiveness of the dyadic intervention on the psychosocial outcomes of children with ID and their caregiving mothers. The qualitative component will consist of longitudinal in-depth interviews with mothers to understand the experiences, perceived changes, and factors that facilitate the process. Art-based assessment will also be used to understand the changes in the emotional expression of children with ID. Data collected will be triangulated to provide an integrative evaluation of the effectiveness of the intervention.

ELIGIBILITY:
Eligible participants are mother-child dyads that fulfill the following inclusion criteria.

* The child is 6-12 years old (primary school student);
* The child is diagnosed with mild to moderate ID, IQ score ranges from 35 to 69 (based on the assessment conducted by certified clinicians);
* By the judgement of the health/school professional staff, the child is capable of responding to assessments and participating in group activities;
* The dyad is willing and able to give consent for participation.

Exclusion Criteria:

* The dyad is currently participating in any other behavioral or pharmacological trial
* Either member of the dyad have other contraindications or severe comorbidities that may impair their full participation (e.g., severe physical disabilities)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only mothers are eligible for this study
Enrollment: 154 (Estimated)
Dates: Start 2022-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Baseline Mothers' Parenting Stress level at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Chinese validated version of the Parenting Stress Index Short-Form will be used to assess the level of parenting stress of the mothers. The index assesses parenting stress in three domains: (i) parental distress, (ii) parent-child dysfunctional interaction, and (iii) difficult child. Higher scores represent higher parenting stress. This index will be filled in by mothers.
Change of Baseline Mothers' Burnout level at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Chinese validated version of the client burnout subscale of the Copenhagen Burnout Inventory will be used to assess the level of burnout of the mothers. Higher scores represent higher burnout. This inventory will be filled in by mothers.
Change of Baseline Mothers' perceive Parent-Child Relationship at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The subscales of parent-child communication and satisfaction with parenting from the Parent-Child Relationship Inventory will be used to assess the mother's perception of the parent-child relationship. Higher scores represent a more positive perception of certain aspects of the parent-child relationship. The research team will undertake the Chinese translation process. This inventory will be filled in by mothers.

SECONDARY OUTCOMES:
Change of Baseline Mothers' Positive and Negative Affect level at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Chinese validated version of the International Positive and Negative Affectivity Schedule - Short Form will be used to assess the level of positive and negative affectivity of mothers. The scale yields two scores indicating the level of positive and negative affect separately. Higher scores represent a higher level of positive or negative affect. This scale will be filled in by mothers.
Change of Baseline Mothers' Quality of Life level at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Hong Kong-Chinese validated version of the WHO Quality of Life Scale brief version will be used to assess the level of quality of life of mothers. Four main domains of Quality of Life will be assessed, including physical, psychological, social relationship, and environmental. Higher scores represent a higher level of quality of life. The scale will be filled in by mothers.
Change of Baseline Mothers' Psychological Well-being at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Hong Kong Cantonese validated version of The World Health Organisation- Five Well-Being Index (WHO-5) will be used to assess the level of psychological well-being of mothers. The scale yields a raw score and will be multiplied by 4 to yield a percentage score. Higher scores represent a higher level of psychological well-being. The scale will be filled in by mothers.
Change of Baseline Children's Mood States at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Ottawa Mood Scales will be adopted to assess the mood states of children with intellectual disabilities. The scale composes of 5 items that assess the level of mood, anger, worry, stress, and self-regulation. Visual clues, such as schematic faces, numerical scales, and thermometer icons, are included for facilitating the understanding. The research team will undertake the Chinese translation process. This inventory will be filled in by children with intellectual disabilities with assistance.
Change of Baseline Children's Emotional Expression at 2 months, 5 months, and 8 months | Baseline, Month 2, Month 5, Month 8
  The Face Stimulus Assessment will be utilized to assess the level of emotional expression of children with intellectual disabilities. The assessment contains a series of three A4-size stimulus drawing templates: the first is a pre-drawn face, the second is a face outline, and the third is a blank sheet of paper. Participants will be asked to use the markers provided on the templates individually. The whole process and the sketches will be assessed through a quantitative and qualitative approach following guidelines from the FSA E-Packet and Rating Manual (2nd ed.)The sketches will also be scanned to analyze the pattern of color usage. This assessment will be filled in by children with intellectual disabilities with assistance.
Change of Baseline Children's Behavioral and Emotional Problem at 2 months, 5 months, | Baseline, Month 2, Month 5, Month 8
  The Hong Kong-Chinese authorized version of the Child Behavior Checklist (Teachers' Report Form) will be used to assess the level of Behavioral and Emotional Problems of children with intellectual disabilities. The checklist yields three scores on externalizing, internalizing, and total behavioral problems, and eight syndromes are withdrawn, somatic complaints, anxious/depressed, thought problems, social problems, attention problems, delinquent behaviors, and aggressive behavior. Higher scores indicate greater manifestations of that area of behavioral and emotional problems. The checklist will be filled in by corresponding teachers or social workers.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre on Behavioral Health HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the principal investigator upon reasonable request. The data are not publicly available due to it involves personal and clinical data from children with intellectual disability and their mothers.
Supporting Information: Study Protocol, ICF
Time Frame: 3 years after the completion of the study
Access Criteria: The principal investigator will review each request and decide if data will be available to other researchers.

REFERENCES:
- [Derived] Lo TLT, Wan AHY, Fong TCT, Wong PKS, Lo HHM, Chan CKP, Ho RTH. Protocol for a mixed-methods randomised controlled trial evaluating the effectiveness of a dyadic expressive arts-based intervention in improving the psychosocial well-being of children with intellectual disability in special schools and their mothers. BMJ Open. 2023 Jul 7;13(7):e067239. doi: 10.1136/bmjopen-2022-067239. PMID 37419633

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT05214859/Prot_SAP_004.pdf